CLINICAL TRIAL: NCT05296382
Title: Relative Bioavailability of Tebipenem (SPR994) Crushed Tablet Formulation Administered by Nasogastric Tube in Healthy Subjects
Brief Title: Bioavailability of Tebipenem (SPR994) Crushed Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HHC-2021-0354
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Relative Bioavailability

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Crushed Tebipenem Tablet with Tube feeds (Experimental): Crushed tebipenem tablets will be administered by syringe through the nasogastric tube and flushed with water to ensure all drug is passed through. Subjects will also receive concurrent enteral tube feeds (feeds run for 2h before dose and 4h post-dose).
  Interventions: Drug: Tebipenem tablet form; Other: Tube feeds
- Whole Tebipenem Tablet (Experimental): Tebipenem tablet will be swallowed whole without crushing.
  Interventions: Drug: Tebipenem tablet form
- Crushed Tebipenem Tablet without Tube feeds (Experimental): Crushed tebipenem tablets will be administered by syringe through the nasogastric tube and flushed with water to ensure all drug is passed through.
  Interventions: Drug: Tebipenem tablet form; Other: Tube feeds

INTERVENTIONS:
Drug: Tebipenem tablet form — Tebipenem tablets will be administered intact or crushed
Other: Tube feeds — Tebipenem tablets will be administered with or without tube feeds
  Arms: Crushed Tebipenem Tablet with Tube feeds; Crushed Tebipenem Tablet without Tube feeds

SUMMARY:
The purpose of this study is to measure the amount of the antibiotic, tebipenem (SPR994) that is bioavailable after crushing the tablet and administering through a feeding tube with and without tube feeds.

DETAILED DESCRIPTION:
This study will enroll 12 healthy volunteers and will take place in the Clinical Research Center at Hartford Hospital. Each volunteer will receive 2 doses (~22h washout period between doses) and will be randomly assigned to three treatment groups:

1) intact tebipenem 600mg dose (2 300mg tablets) taken orally; 2) a crushed tebipenem 600mg dose (2 300mg tablets) suspended in water and administered via the NGT; 3) a crushed tebipenem 600mg dose (2 300mg tablets) suspended in water and administered via a nasogastric tube with concurrent enteral tube feeds (run for 2h before dose and 4h post-dose). Crushed tablets will be administered by syringe through the nasogastric tube. An additional 150ml of water will be used to rinse out any remaining drug in syringe and administered to the volunteers to ensure delivery of the entire dose.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the trial, give written informed consent, and comply with the trial restrictions.
2. Gender: male or female with a negative serum pregnancy test (β-human chorionic gonadotropin) at Screening and Day -1; females may be of childbearing potential or of non-childbearing potential.
3. Age >= 18 years at screening

Exclusion Criteria:

1. Female who is pregnant, lactating, or at risk of becoming pregnant during this trial.
2. History of hypersensitivity or allergy to tebipenem or its derivatives and any β-lactam antibiotic.
3. History of hypersensitivity to lidocaine or lidocaine derivatives.
4. Concurrently receiving sodium valproic acid or valproate derivatives.
5. Concurrently receiving probenecid.
6. Body Mass Index (BMI) ≥ 35 kg/m2
7. Creatinine clearance (CrCl) < 50ml/min, as calculated by Cockcroft-Gault using ideal body weight
8. Presence of anemia, thrombocytopenia, or leukopenia as defined by hematocrit, platelet, or white blood cell count < 75% of the lower limit of normal
9. Aspartate transaminase, alanine aminotransferase, or alkaline phosphatase greater than five times upper limit of normal.
10. Total bilirubin greater than three times the upper limit of normal.
11. Any known active co-morbidity listed on medical history i.e., seizures or that becomes apparent during physical examination.
12. Positive urine drug screen (cocaine, Tetrahydrocannabinol, opiates, benzodiazepines, and amphetamines).
13. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
14. Use of tobacco- or nicotine-containing products in excess of the equivalence of 5 cigarettes per day.
15. Consumption of caffeine within 3 days of the study.
16. Use of prescription or nonprescription drugs, vitamins, or dietary supplements within 7 days or 5 half-lives, whichever is longer (with the exception of acetaminophen at doses of ≤ 1 g/day). The use of hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine devices, post-coital contraceptive methods) is permitted.
17. Males who are not surgically sterilized (with female partners of childbearing potential) and females of childbearing potential who do not agree to use two highly effective methods of contraception from screening, during this trial, and for 90 days after the last dose of study drug.
18. History or current presence of nasal structural abnormalities including a broken nose or deviated septum.
19. Employee of the Center for Anti-Infective Research and Development, Clinical Research Center, or the Sponsor.
20. Any other documented reason felt by the investigator to potentially affect the outcomes of the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Tebipenem drug exposure | 8 hours
  Tebipenem total and free blood concentrations following the tebipenem dose (intact)
Tebipenem drug exposure | 8 hours
  Tebipenem total and free blood concentrations following the tebipenem dose (crushed and administered via NGT)
Tebipenem drug exposure | 8 hours
  Tebipenem total and free blood concentrations following the tebipenem dose (crushed and administered with tube feeds via NGT)

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States